CLINICAL TRIAL: NCT05029934
Title: Efficacy of EndoClot™ Spraying After Endoscopic Resection of Large Colorectal Polyps: A Randomized Trial.
Brief Title: Efficacy of EndoClot™ Spraying After Endoscopic Resection of Large Colorectal Polyps
Acronym: EndoClot™
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment of study patients
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PV7200
Record Dates: First submitted 2021-08-29; First posted 2021-09-01 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Wound Endoscopical, Colon; After Polyp Resection, Colon
Keywords: colon endoscopic mucosa resection (EMR); delayed bleeding; colonoscopy; polyp resection

STUDY DESIGN:
Intervention Model Description: use of EndoClot adhesive after resection vs no use of any preventive action against delayed bleeding (control group)
Who Masked: Participant
Masking Description: Patients will not be informed about the use of EndoClot adhesive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EndoClot group (Active Comparator): patients who are being provided with EndoClot adhesive spray after polyp resection
  Interventions: Procedure: use of EndoClot
- Control group (Sham Comparator): no further prophylactic bleeding prevention after polyp resection
  Interventions: Procedure: use of EndoClot

INTERVENTIONS:
Procedure: use of EndoClot — deployment of EndoClot adhesive spray

SUMMARY:
The effectiveness of colonoscopy in reducing colorectal cancer mortality relies on the detection and removal of neoplastic polyps. Effective and safe resection of larger polyps is particularly important due to their higher potential of malignancy. Large polyps ≥20mm are removed by so-called endoscopic mucosal resection (EMR) (and occasionally endoscopic submucosal dissection (ESD)) using electrocautery snares. Resection of these large polyps is associated with a risk of severe complications that may require hospitalization and additional interventions. The most common risk is delayed bleeding which is observed in approximately 2-10% of patients. In a recent randomized trial, clipping has been shown to reduce bleeding esp. on the right colonic side. However, clipping of larger areas is time consuming and may add to costs in several ways.

Our primary aim is to examine whether EndoClot™ application (a special form of longer lasting spray on the mucosal defect after EMR/ESD of large non-pedunculated colorectal polyps (≥20mm) will reduce the risk of delayed bleeding. We hypothesize that EndoClot™ application will reduce the risk of delayed bleeding by at least 3/4 (i.e. from 7.5% to 1.5%) based on an initial assumption of a 7.5% delayed bleeding rate.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common cause of cancer death in the United States and Europe. The effectiveness of colonoscopy in reducing the risk of dying from colorectal cancer relies on the detection and safe resection of neoplastic polyps to prevent incident cancers. Most polyps are small and can be easily removed using snare with or without electrocautery. Because the risk of prevalent cancer or transition to cancer increases with polyp size, effective and safe resection of large polyps is particularly important.

Endoscopic mucosal resection (EMR) is evolving as the primary endoscopic technique to remove large non-pedunculated polyps. These flat or sessile polyps are defined as lateral spreading tumors with a low vertical axis that extend laterally along the luminal wall. Several mostly retrospective studies from Europe, the U.S. and Japan, have demonstrated a high "cure" rate, with results lending credence to the shift from surgical resection to endoscopic management of these lesions. Of concern, however, is 1) a fairly high overall complication rate of 8-26% in prospective studies3-7, and 2) as well the persistence of residual neoplasia on follow-up endoscopy ranging from 16% to 46%3, 6, 8. The former is the main topic of the present study.

Severe complications including bleeding associated with a standard diagnostic or screening colonoscopy, which may include resection of predominantly smaller polyps, are uncommon. Significant bleeding occurs in 0.2 to 0.5% of patients (defined as a 2mg drop in Hemoglobin) 9, 10. The risk of severe complications increases with polyp size; here, again, the most common complication is bleeding reported in 2 to 24% of polyp resections. In one recent analysis the rate of delayed bleeding in colonic EMR was 7.5%1.

In addition to size, other factors may affect complications. These include type of resection (piecemeal versus en-bloc), polyp location (right colon with a thinner wall than the left colon), age and comorbidities, especially those that affect clotting abilities (e.g. renal insufficiency, liver disease, use of anticoagulation). Studies that have examined variables, which may directly decrease the risk of complications associated with large polyp resection, are limited.

It is apparent that resection of a large polyp leaves behind a large mucosal defect. The mucosal ulcer that forms after polyp resection can take several weeks to heal. Bleeding complications typically occur within 7 to 10 days, requiring often admission, a repeat colonoscopy to stop bleeding, and possible blood transfusions. The rates depend on size, and have been shown to be around 1.5%-2.6% overall. It is significantly higher in larger adenomas of 2 cm and more, namely 6.5% in another recent meta analysis.

To reduce the risk of bleeding various measures have been proposed which also have been summarized in several recent meta analyses. These include coagulation, clipping and others, but only few randomized trials are available: Coagulation not effective in a recent meta analysis14, but only 4 of the 12 studies were randomized and these included all mostly smaller polyps or polyps of all sizes or pedunculated polyps. In a recent randomized trial, clipping has been shown to reduce bleeding esp. on the right colonic side. However, clipping of larger areas is time consuming and may add to costs in several ways.

Our primary aim is to examine whether EndoClot™ application (a special form of longer lasting spray on the mucosal defect after EMR/ESD of large non-pedunculated colorectal polyps (≥20mm) will reduce the risk of delayed bleeding. We hypothesize that EndoClot™ application will reduce the risk of delayed bleeding by at least 3/4 (i.e. from 7.5% to 1.5%) based on an initial assumption of a 7.5% delayed bleeding rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a ≥20mm colon non-pedunculated polyp who are undergoing an ESD or EMR resection
* signed Informed Consent

Exclusion Criteria:

* Patients with known (biopsy proven) or strongly suspected invasive carcinoma in a potential study polyp
* Pedunculated polyps (as defined by Paris Classification type Ip or Isp)
* ulcerated depressed lesions (as defined by Paris Classification type III)
* polyposis syndromes
* inflammatory bowel disease
* emergency colonoscopy
* Poor general health (ASA (American Society of Anaesthesiologists) class>3)
* Patients with coagulopathy with an elevated International Normalized Ratio (INR )≥1.5, or platelets <50
* Poor bowel preparation
* pregnancy or breastfeeding
* Intervention planned using ORISE™ (Boston Medical) or LIFTUP™ (Ovesco) as lifting agents

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
delayed bleeding complication: hospitalization | 30 days
  hospitalization after subsequent return to unit / health care facility for evaluation of rectal bleeding
delayed bleeding complication: transfusion | 30 days
  a patient who subsequently had to return to the unit and/or any health care facility for evaluation of rectal bleeding AND who required transfusion
delayed bleeding complication: repeat endoscopy | 30 days
  a patient who subsequently had to return to the unit and/or any health care facility for evaluation of rectal bleeding AND who required a repeat colonoscopy or sigmoidoscopy for examination of the polypectomy site or control of bleeding
delayed bleeding complication: | 30 days
  a patient who subsequently had to return to the unit and/or any health care facility for evaluation of rectal bleeding AND who required surgery

SECONDARY OUTCOMES:
Technical handling | 20 minutes (assumed deployment time)
  product deployment assumed quantity of entire vial: < 50%/50-70%/100%
Overall complications | procedure to day 30
  an aggregate of all complications that occur at the time of the procedure or during follow-up
Factors associated with complications: polyp size | 30 days
  Factors that may be associated with complications, esp. bleeding
Factors associated with complications: polyp location | 30 days
  Factors that may be associated with complications, esp. bleeding: location of the polyp in the colon (right, left, rectum)
Factors associated with complications: polyp histology | 30 days
  Factors that may be associated with complications, esp. bleeding
Factors associated with complications: polyp morphology | 30 days
  Factors that may be associated with complications, esp. bleeding
Factors associated with complications: polyp resection time | 30 days
  Factors that may be associated with complications, esp. bleeding

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Vivantes Auguste-Viktoria-Klinikum, Berlin
  - University Hospital Hamburg Eppendorf, Hamburg
  - Evangelisches Amalie Sieveking Krankenhaus, Hamburg
  - UKGM Marburg, Klinik für Gastroenterologie, Marburg
  - Klinikum Südstadt Rostock, Rostock

REFERENCES:
- [Background] Pohl H, Grimm IS, Moyer MT, Hasan MK, Pleskow D, Elmunzer BJ, Khashab MA, Sanaei O, Al-Kawas FH, Gordon SR, Mathew A, Levenick JM, Aslanian HR, Antaki F, von Renteln D, Crockett SD, Rastogi A, Gill JA, Law RJ, Elias PA, Pellise M, Wallace MB, Mackenzie TA, Rex DK. Clip Closure Prevents Bleeding After Endoscopic Resection of Large Colon Polyps in a Randomized Trial. Gastroenterology. 2019 Oct;157(4):977-984.e3. doi: 10.1053/j.gastro.2019.03.019. Epub 2019 Mar 15. PMID 30885778
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Brooker JC, Saunders BP, Shah SG, Thapar CJ, Suzuki N, Williams CB. Treatment with argon plasma coagulation reduces recurrence after piecemeal resection of large sessile colonic polyps: a randomized trial and recommendations. Gastrointest Endosc. 2002 Mar;55(3):371-5. doi: 10.1067/mge.2002.121597. PMID 11868011
- [Background] Conio M, Repici A, Demarquay JF, Blanchi S, Dumas R, Filiberti R. EMR of large sessile colorectal polyps. Gastrointest Endosc. 2004 Aug;60(2):234-41. doi: 10.1016/s0016-5107(04)01567-6. PMID 15278051
- [Background] Ferrara F, Luigiano C, Ghersi S, Fabbri C, Bassi M, Landi P, Polifemo AM, Billi P, Cennamo V, Consolo P, Alibrandi A, D'Imperio N. Efficacy, safety and outcomes of 'inject and cut' endoscopic mucosal resection for large sessile and flat colorectal polyps. Digestion. 2010;82(4):213-20. doi: 10.1159/000284397. Epub 2010 Jun 24. PMID 20588036
- [Background] Moss A, Bourke MJ, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Chen RY, Byth K. Endoscopic mucosal resection outcomes and prediction of submucosal cancer from advanced colonic mucosal neoplasia. Gastroenterology. 2011 Jun;140(7):1909-18. doi: 10.1053/j.gastro.2011.02.062. Epub 2011 Mar 8. PMID 21392504
- [Background] Swan MP, Bourke MJ, Alexander S, Moss A, Williams SJ. Large refractory colonic polyps: is it time to change our practice? A prospective study of the clinical and economic impact of a tertiary referral colonic mucosal resection and polypectomy service (with videos). Gastrointest Endosc. 2009 Dec;70(6):1128-36. doi: 10.1016/j.gie.2009.05.039. Epub 2009 Sep 12. PMID 19748615
- [Background] Arebi N, Swain D, Suzuki N, Fraser C, Price A, Saunders BP. Endoscopic mucosal resection of 161 cases of large sessile or flat colorectal polyps. Scand J Gastroenterol. 2007 Jul;42(7):859-66. doi: 10.1080/00365520601137280. PMID 17558911
- [Background] Levin TR, Zhao W, Conell C, Seeff LC, Manninen DL, Shapiro JA, Schulman J. Complications of colonoscopy in an integrated health care delivery system. Ann Intern Med. 2006 Dec 19;145(12):880-6. doi: 10.7326/0003-4819-145-12-200612190-00004. PMID 17179057
- [Background] Ko CW, Riffle S, Michaels L, Morris C, Holub J, Shapiro JA, Ciol MA, Kimmey MB, Seeff LC, Lieberman D. Serious complications within 30 days of screening and surveillance colonoscopy are uncommon. Clin Gastroenterol Hepatol. 2010 Feb;8(2):166-73. doi: 10.1016/j.cgh.2009.10.007. Epub 2009 Oct 20. PMID 19850154
- [Background] Reumkens A, Rondagh EJ, Bakker CM, Winkens B, Masclee AA, Sanduleanu S. Post-Colonoscopy Complications: A Systematic Review, Time Trends, and Meta-Analysis of Population-Based Studies. Am J Gastroenterol. 2016 Aug;111(8):1092-101. doi: 10.1038/ajg.2016.234. Epub 2016 Jun 14. PMID 27296945
- [Background] Jaruvongvanich V, Prasitlumkum N, Assavapongpaiboon B, Suchartlikitwong S, Sanguankeo A, Upala S. Risk factors for delayed colonic post-polypectomy bleeding: a systematic review and meta-analysis. Int J Colorectal Dis. 2017 Oct;32(10):1399-1406. doi: 10.1007/s00384-017-2870-0. Epub 2017 Aug 5. PMID 28779355
- [Background] Hassan C, Repici A, Sharma P, Correale L, Zullo A, Bretthauer M, Senore C, Spada C, Bellisario C, Bhandari P, Rex DK. Efficacy and safety of endoscopic resection of large colorectal polyps: a systematic review and meta-analysis. Gut. 2016 May;65(5):806-20. doi: 10.1136/gutjnl-2014-308481. Epub 2015 Feb 13. PMID 25681402
- [Background] Boumitri C, Mir FA, Ashraf I, Matteson-Kome ML, Nguyen DL, Puli SR, Bechtold ML. Prophylactic clipping and post-polypectomy bleeding: a meta-analysis and systematic review. Ann Gastroenterol. 2016 Oct-Dec;29(4):502-508. doi: 10.20524/aog.2016.0075. Epub 2016 Jul 28. PMID 27708518
- [Background] ASGE Standards of Practice Committee; Anderson MA, Ben-Menachem T, Gan SI, Appalaneni V, Banerjee S, Cash BD, Fisher L, Harrison ME, Fanelli RD, Fukami N, Ikenberry SO, Jain R, Khan K, Krinsky ML, Lichtenstein DR, Maple JT, Shen B, Strohmeyer L, Baron T, Dominitz JA. Management of antithrombotic agents for endoscopic procedures. Gastrointest Endosc. 2009 Dec;70(6):1060-70. doi: 10.1016/j.gie.2009.09.040. Epub 2009 Nov 3. No abstract available. PMID 19889407
- [Background] Karita M, Tada M, Okita K, Kodama T. Endoscopic therapy for early colon cancer: the strip biopsy resection technique. Gastrointest Endosc. 1991 Mar-Apr;37(2):128-32. doi: 10.1016/s0016-5107(91)70669-x. PMID 2032596
- [Background] Tullavardhana T, Akranurakkul P, Ungkitphaiboon W, Songtish D. Efficacy of submucosal epinephrine injection for the prevention of postpolypectomy bleeding: A meta-analysis of randomized controlled studies. Ann Med Surg (Lond). 2017 Jun 6;19:65-73. doi: 10.1016/j.amsu.2017.05.035. eCollection 2017 Jul. PMID 28652912
- [Background] Klein A, Tate DJ, Jayasekeran V, Hourigan L, Singh R, Brown G, Bahin FF, Burgess N, Williams SJ, Lee E, Sidhu M, Byth K, Bourke MJ. Thermal Ablation of Mucosal Defect Margins Reduces Adenoma Recurrence After Colonic Endoscopic Mucosal Resection. Gastroenterology. 2019 Feb;156(3):604-613.e3. doi: 10.1053/j.gastro.2018.10.003. Epub 2018 Oct 6. PMID 30296436